CLINICAL TRIAL: NCT02651402
Title: A Hybrid Effectiveness-Implementation Trial of Group Cognitive Behavior Therapy (CBT) in Urban Schools
Brief Title: A Hybrid Effectiveness-Implementation Trial of Group CBT in Urban Schools
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: University of Pennsylvania (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 15-012311; 1R01MH108555-01 (NIH)
Record Dates: First submitted 2016-01-07; First posted 2016-01-11 (Estimated); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Anxiety Disorders
Keywords: Anxiety Disorders; Internalizing; Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- FRIENDS for Life Train-the-Trainer (Active Comparator): Therapists implement FRIENDS (a CBT protocol for students with anxiety) in the school setting, while supported by their supervisor assigned to the Train-the-Trainer (TT) implementation strategy (supervisors participate in training workshops on conducting supervision with active therapists).
  Interventions: Behavioral: FRIENDS for Life; Behavioral: Train-the-Trainer
- Adapted FRIENDS Train-the-Trainer (Experimental): Therapists implement an adapted version of FRIENDS (aFRIENDS) in the school setting while supported by their supervisor assigned to the TT strategy.
  Interventions: Behavioral: Adapted FRIENDS; Behavioral: Train-the-Trainer
- Adapted FRIENDS Train-the-Trainer Plus (Experimental): Therapists implement aFRIENDS in the school setting while supported by their supervisor assigned to the Train-the-Trainer Plus (TT+) implementation strategy (supervisors participate in training workshops and receive further/on-going consultation on conducting supervision with active therapists).
  Interventions: Behavioral: Adapted FRIENDS; Behavioral: Train-the-Trainer Plus

INTERVENTIONS:
Behavioral: FRIENDS for Life — Friends for Life (FRIENDS): FRIENDS, a GCBT program, is an effective program for the prevention and treatment of anxiety disorders in children evidenced by a meta-analysis on school-based interventions for at-risk and clinically anxious youth. FRIENDS was developed based on the view that anxiety is a tripartite construct involving physiological, cognitive, and behavioral components. Core Intervention components: Experts in CBT for childhood anxiety disorders have identified 5 essential components: psychoeducation, somatic management skills training, cognitive restructuring, exposure methods, and contingency management. The FRIENDS protocol consists of 10 weekly sessions and two booster sessions. We included the booster sessions in the regular protocol for a total of 12 sessions.
  Other Names: FRIENDS
  Arms: FRIENDS for Life Train-the-Trainer
Behavioral: Adapted FRIENDS — Adapted Friends (aFRIENDS): We conducted planned adaptations to the FRIENDS protocol based on our collective experience with the protocol and qualitative data (focus group and interviews). We followed procedures developed by Lee and colleagues, including surveying service providers and trainers regarding the appropriateness of FRIENDS for the target population. Changes were made to the language (idioms, metaphors, words), cultural fit (cultural values), methods (session length, number of sessions), activities (in-session practices), which resulted in additions and substitutions in these areas while maintaining the 5 essential components of the treatment. aFRIENDS is a briefer (8-session) and more engaging and culturally-sensitive protocol than FRIENDS.
  Other Names: aFRIENDS
  Arms: Adapted FRIENDS Train-the-Trainer; Adapted FRIENDS Train-the-Trainer Plus
Behavioral: Train-the-Trainer — Train the Trainer (TT): agency supervisors are trained to conduct effective supervision (one initial training and 2 booster sessions), and then go on to train intervention therapists.
  Other Names: TT
  Arms: Adapted FRIENDS Train-the-Trainer; FRIENDS for Life Train-the-Trainer
Behavioral: Train-the-Trainer Plus — Train the Trainer Plus (TT+): a modified train-the-trainer approach by which supervisors receive training plus extended on-going consultation on conducting effective supervision with intervention therapists.
  Other Names: TT+
  Arms: Adapted FRIENDS Train-the-Trainer Plus

SUMMARY:
Unresolved psychological problems, such as anxiety, affect a significant number of our students and interfere with their ability to attend, actively participate, and prosper in school. This project will expand the capacity of selected mental health agencies to provide services in the participating schools through school therapeutic services (STS). The project will provide enhanced training in evidence-based behavioral health interventions to school-based mental health providers. The services will be implemented by STS Bachelor's or Master's level therapists supervised by their mental health agency supervisors (Internal Support), who are in turn supported by the research team (Train-the-Trainer) or external consultants (Train the Trainer+).

DETAILED DESCRIPTION:
Background/Purpose: This project will expand the capacity of selected mental health agencies to provide services in the participating schools through school therapeutic services (STS). The project will provide enhanced training in evidence-based behavioral health interventions to school-based mental health providers. The services will be implemented by STS Master's level therapists supervised by their mental health agency supervisors (Internal Support), who are in turn supported by the research team (TT) or external consultants (TT+).

Population: 18 schools in Philadelphia will be chosen for participation. Students who present excessive anxiety in grades 4-8 would be potentially eligible to participate in the interventions offered by the agencies' therapists in their school.

Intervention: This study is designed to test: a) the effectiveness of an adapted version of a group cognitive behavioral therapy program (aFRIENDS) compared to the original version of this program (FRIENDS), and b) the effectiveness of two implementation support strategies for aFRIENDS: Train-the-Trainer and Train-the-Trainer Plus. aFRIENDS is a shorter, more culturally sensitive, focused, and feasible CBT for anxiety in children than FRIENDS and addresses one of the major barriers to implementation (intervention-context fit).

Design: Therapists and supervisors will be randomly assigned to one of three conditions: a) FRIENDS with Train-the-Trainer implementation strategy (i.e., Masters-level supervisors receive training by experts on conducting supervision); b) aFRIENDS with Train-the-Trainer strategy; c) aFRIENDS using the Train-the-Trainer Plus strategy (i.e., supervisors receive training and consultation by experts on conducting supervision).

Analyses: Effectiveness will be measured by comparing A to B; Implementation will be measured by comparing B to C. Agency therapists will conduct all treatment groups in the schools.

ELIGIBILITY:
Inclusion Criteria:

1. Supervisors: Any participating agency clinical supervisor with a Master's degree or higher in a mental health field.
2. Therapists: Any STS therapist with a Bachelor's degree or higher who provides services in one of the 18 participating schools.
3. Students: Any student enrolled in grades 4-8 in one of the participating schools, who had been referred to the STS program in their school and who meets study screening and diagnostic criteria. The screening criterion is a Total score > 25 on Screen for Child Anxiety Related Disorders (SCARED) completed by a parent or school staff member. This student must also present a primary positive or intermediate diagnosis of Separation Anxiety Disorder (SAD]) Generalized Anxiety Disorder (GAD), or Social Phobia (SP) on the Anxiety Disorders Interview Schedule (ADIS); completed by a parent during the eligibility evaluation.
4. If, at the conclusion of the eligibility evaluation, students do not meet diagnostic criteria (see above) to participate in the study, but parents and school staff continue to express concern about functional impairment, students will be permitted to participate in the intervention sessions (with parent permission). We also expect that there might be a very small number of eligible children whose parents may not give consent, and some of these parents and school personnel might want these children to benefit from the intervention. As such, we would like to offer these children the opportunity to participate along with the research subjects. This group of students will not be identified as "research subjects" and study data will not be collected from them. However, parents will be asked to sign a permission form for the video recording of the group sessions. This is the procedure we currently follow for our National Institute of Child Health and Human Development (NICHD) funded project, which has been approved by the Institutional Review Board (IRB) of The Children's Hospital of Philadelphia and School District of Philadelphia.

Exclusion Criteria:

1. Supervisors or therapists not involved in STS.
2. Students with Special Education classification of "Intellectual Disability;" children whose primary diagnosis is not SAD, GAS or SP.
3. Students with a history of psychotic or autistic spectrum disorders according to school records.

   * Students meeting criteria in #2 & #3 above will be excluded from participation because they would be unlikely to benefit from Global Cognitive Behavioral Therapy (GCBTS).

Subjects that do not meet all of the enrollment criteria may not be enrolled. Any violations of these criteria must be reported in accordance with IRB Policies and Procedures.

Ages: 8 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 495 (Actual)
Dates: Start 2016-02; Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Change in Manifest Anxiety Scale for Children (MASC) from Baseline to Post Intervention completed by parents and children | Up to 12 weeks
  Effectiveness between treatment groups will be assessed by comparing the change in diagnostic status from pre to post intervention. Diagnostic status will be assessed using the Anxiety Disorders Interview Schedule for Children (ADIS-P) which includes a semi-structured interview used to determine diagnostic status and outcome. Clinical judgement is used to generate a Clinician Severity Rating (CSR). A CSR >4 is a clinical diagnosis of an anxiety disorder, CSR=3 patient at risk for developing a disorder.

SECONDARY OUTCOMES:
Cost Effectiveness | Duration of Project (5 years)
  A Cost Benefit Analysis will be conducted across both interventions and implementation strategies, comparing material expenses, personnel effort, agency and school district salaries, etc.

OTHER OUTCOMES:
Implementation Fidelity: Train-the-Trainer (TT) to Train-the-Trainer Plus (TT+) for the implementation of aFRIENDS. | Duration of Project (5 years)
  Using fidelity checklists, the ability of therapists to implement the interventions (as clinically intended), will be measured and compared across support implementation support strategies (TT vs. TT+).

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo B Eiraldi, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Eiraldi R, Lawson GM, Glick HA, Khanna MS, Beidas R, Fishman J, Rabenau-McDonnell Q, Wilson T, Comly R, Schwartz BS, Jawad AF. Implementation fidelity, student outcomes, and cost-effectiveness of train-the-trainer strategies for Masters-level therapists in urban schools: results from a cluster randomized trial. Implement Sci. 2024 Jan 25;19(1):4. doi: 10.1186/s13012-023-01333-9. PMID 38273369
- [Derived] Lawson GM, Comly R, Beidas RS, Khanna MS, Goldstein J, Brizzolara-Dove S, Wilson T, Rabenau-McDonnell Q, Eiraldi R. Therapist and supervisor perspectives about two train-the-trainer implementation strategies in schools: A qualitative study. Implement Res Pract. 2023 Aug 3;4:26334895231190854. doi: 10.1177/26334895231190854. eCollection 2023 Jan-Dec. PMID 37790186
- [Derived] Eiraldi R, Khanna MS, Jawad AF, Fishman J, Glick HA, Schwartz BS, Cacia J, Wandersman A, Beidas R. A hybrid effectiveness-implementation cluster randomized trial of group CBT for anxiety in urban schools: rationale, design, and methods. Implement Sci. 2016 Jul 12;11:92. doi: 10.1186/s13012-016-0453-z. PMID 27405587

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-05): https://cdn.clinicaltrials.gov/large-docs/02/NCT02651402/Prot_SAP_000.pdf